CLINICAL TRIAL: NCT06071234
Title: An Exploration of 3D Reconstruction Tool for Preoperative Evaluation in Reducing Ischemic Complications of Flap and Nipple-Areolar Complex (NAC) After Nipple-sparing Mastectomy
Brief Title: Preoperative Evaluation of 3D Reconstruction Tool for Nipple-sparing Mastectomy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Kun Wang, Professor, Guangdong Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3D-RECON
Record Dates: First submitted 2023-10-03; First posted 2023-10-06 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D-reconstruction group (Experimental): The participant's breast blood supply was assessed preoperatively using 3D reconstruction technology, and the flap was separated intraoperatively using a combination of electrocautery and sharp dissection.
  Interventions: Procedure: 3D reconstruction technology
- Normal group (Active Comparator): Participants are not evaluated preoperatively using 3D reconstruction technology and flap separation is performed using electrosurgical knife intraoperatively.
  Interventions: Procedure: 3D reconstruction technology

INTERVENTIONS:
Procedure: 3D reconstruction technology — Preoperative application of 3D reconstruction technology to evaluate the breast blood supply of participants and observe whether the incidence of ischemic complications in the flap and nipple areola complex is reduced compared to surgery without preoperative evaluation.

SUMMARY:
The goal of this clinical study is to explore whether preoperative application of 3D reconstruction tool can reduce the occurrence of ischemic complications in the flap and nipple areola complex after surgery.

DETAILED DESCRIPTION:
The 3D reconstruction tool was applied preoperatively to assess the blood supply and volume of participants' breasts and to recommend personalized prosthesis volume. Compared with electrosurgical knife separation，the flap was separated intraoperatively using a combination of cold knife and electrosurgical knife to observe whether there was a difference in the incidence of ischemic complications of participants' nipple areola complex and flap, and whether the use of the 3D tool in the preoperative assessment was effective in reducing the occurrence of postoperative ischemic complications.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed diagnosis of breast cancer
* Age: 18 to 70 years old
* No infiltration of the nipple-areola complex and negative histopathology of the nipple basal margins;
* Participants who meet the indications for breast conserving surgery require total mastectomy and reconstruction;

Exclusion Criteria:

* Inability to tolerate surgery or subjective desire not to undergo nipple-sparing mastectomy;
* Participants with clinical or imaging evidence of preoperative involvement of the nipple/areolar region, including Paget's disease, nipple spillage, inflammatory breast cancer, and/or imaging findings suggesting malignant involvement of the nipple or subareolar tissues, according to the 2023 NCCN guideline recommendations, where retaining the NAC fails to yield negative margins;

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2023-10-08 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Ischemic complications of flap and nipple areola complex | 1 week and 2 week after surgery
  The incidence of ischemic complications in the skin flap and nipple areola complex after NSM surgery

SECONDARY OUTCOMES:
Severity of ischemic complications in the flap and nipple areola complex | 1 week and 2 week after surgery
  Severity of ischemic complications in the skin flap and nipple areola complex after NSM surgery
Duration of surgery | postoperative
  Record the duration of the procedure from the beginning of the incision to the end of the closure of the skin.
Blood loss | Preoperative and 2 hours postoperatively
  Comparison of hemoglobin values in the preoperative blood test with the results of 2-h postoperative test
Breast-Q Satisfaction | Preoperative, 3 months and 1 year postoperatively
  The outcome will be the score (continuous variable ranging from 0 to 100 for linear regression or ordinal categories, ranging from 1 to 4 for ordinallogistic regression, where 1 represents lowest satisfaction and 4 represents highest satisfaction), and the primary predictor of interest will be type of consultation provided.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China